CLINICAL TRIAL: NCT06928402
Title: Comparison of Airway Ultrasound Measurements With Conventional Parameters in Predicting Difficult Intubation
Brief Title: Comparison of Airway Ultrasound Measurements
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Munire BABAYIGIT, Assoc. Prof., Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: SK001
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Intubation; Difficult or Failed
Keywords: airway management; airway ultrasound; difficult intubation; difficult ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway Measurement Group: As this study is observational in nature, no interventions will be performed by the research team. The study will ,nvolve a single group, within which the incidence and prevalence of the outcomes will be assessed.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no interventions will be performed by the research team

SUMMARY:
Evaluating the success of measurements taken with ultrasound airway imaging in predicting difficult intubation by comparing conventional parameters in terms of difficult intubation and the proportion of patients encountered during intubation and characterised as difficult.

DETAILED DESCRIPTION:
Clinical screening tests, which have long been routinely used for airway assessment, do not have sufficient sensitivity and specificity to detect difficult laryngoscopy. The Cormack-Lehane laryngoscopy classification, which can be assessed during direct laryngoscopy, is an invasive procedure and is not suitable for routine preoperative airway assessment. Preoperative airway assessment using ultrasound can help to predict a difficult laryngoscopy and/or difficult intubation and is growing in popularity as a non-invasive diagnostic tool. Several recent studies have emphasised the importance of various ultrasound-mediated airway measurements in predicting difficult intubation, and have shown that measurements with different parameters and data obtained by ratioing some measurements to each other may have an important role. However, the parameters obtained by ultrasound-mediated airway measurement can help determine airway anatomy and guide airway interventions with dynamic real-time images.

In this study, investigators used hyoid bone visibility obtained through preoperative ultrasound evaluation of the upper airway, followed by measurements of the skin-hyoid distance, skin-cricothyroid membrane distance and length, and hyomental distance in two different positions-neutral and extension. The ratios of these measurements were analyzed to predict difficult intubation. Traditional parameters commonly used as indicators of difficult ventilation and/or intubation, such as the Mallampati-Samsoon classification, upper lip bite test, thyromental distance, sternomental distance, neck circumference, maximum mouth opening, Wilson difficult intubation score, and Han ventilation scale, were also included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be operated with endotracheal intubation under elective conditions
* Voluntary patients whose informed consent was obtained,
* Patients older than 18 years
* Patients evaluated in the 1-2-3 category of the American Society of Anaesthesiologist (ASA)

Exclusion Criteria:

* Patients with a history of difficult intubation
* Pregnant patients
* Patients with a history of surgery in the head and neck region
* Patients with a history of trauma or tumour in the head and neck region
* Presence of a syndrome that will cause difficult intubation
* Uncooperative patients,
* Patients with missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases that meet the inclusion and exclusion criteria will be included in the study. Patients will be taken to the operating room after being preoperatively evaluated in the observation room. The patient's anesthetic management will be provided by another anesthesiologist who is not participating in the study and is responsible for the patient. Intraoperative data will be obtained from the patient's anaesthesia follow-up form and the records of the anaesthesia machine. This group will include patients who will be intubated and operated on under general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Ratio of ultrasound-derived parameters with conventional parameters | 1 hour peroperatively
  ultrasound derived parameters: hyoid bone visibility, skin-hyoid distance, skin-hyoid distance, skin-crricothyroid membrane distance, cricothyroid membrane length and hyomental distance measured in neutral and extension and the ratio of these values.
  Conventional parameters: thyromental distance, sternomental distance, upper lip bite test, head-neck movement, presence of retrognathia, neck circumference, maximum mouth opening, Wilson difficult intubation score, Han scale and Mallampati score

SECONDARY OUTCOMES:
Incidence of difficult intubation | 1 hour peroperatively
  Defined as ≥3 intubation attempts by an experienced anesthesiologist, use of adjunctive devices (e.g., stylet, LMA, video laryngoscope), or duration >10 minutes.
Incidence of difficult ventilation | 1 hour preoperatively
  Grade 3 and 4 for Han scale.( Difficulty of mask ventilation (DMV) has been classified using the Han scale.)

CONTACTS AND LOCATIONS:
Overall Officials: Münire Babayiğit, MD, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Ataturk Sanatorium Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No